CLINICAL TRIAL: NCT03754478
Title: Follow-Up of Fitness in Overweight Patients Treated With Physical Activity
Acronym: FUFPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Lausanne (Other)
Collaborators: Hôpital intercantonal de la Broye, Estavayer-le-lac, Switzerland (Unknown)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor Luc Tappy, University of Lausanne
Other Study IDs: 2018-00147
Record Dates: First submitted 2018-10-17; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Exercise Training; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- overweight subjects: Overweight male and females referred to a physical activity program by their primary care physician Intervention is being included in a 3-month physical activity training program
  Interventions: Other: Physical activity training

INTERVENTIONS:
Other: Physical activity training — subjects will enter a 3-month supervised physical activity program during which they will take part to supervised and unsupervised physical activity sessions. Type of physical activity will be selected among a number of available activities (aquagym, aerobics, resistance training, outdoors activities) based on individual needs and preferences); it will consist in 2 weekly supervised activity sessions during which participants will be instructed by a specialist in adapted physical activity, and 2-3 weekly session of unsupervised physical activity which will be performed according to detailed instructions regarding intensity and duration.

SUMMARY:
Although there is increasing evidence that low physical fitness is a risk factor for many non-communicable diseases, the early identification of subjects at risk remains inadequate due to the absence of clear anamnestic and clinical criteria. Defining physical fitness. For the same reason, the monitoring of subjects following lifestyle interventions remains suboptimal.

The aim of this study is to develop a simple field tool to non-invasively assess global physical fitness in overweight patients participating to a physical activity program.

Male and female overweight subjects referred to a physical activity intervention by their primary care physician will be included. Within this program, they will take part to 2 weekly supervised activity sessions during which participants will be instructed by a specialist in adapted physical activity, and 2-3 weekly session of unsupervised physical activity which will be performed according to detailed instructions regarding intensity and duration. In addition, participants will take part to teaching sessions in group of 4-6 patients, addressing the effects of physical activity on metabolism, contra-indications to physical activity, self-monitoring of exercise, and prevention of injuries Their physical fitness will be assessed at inclusion (ie before starting the exercise program) and at the end of the 3-month program. This will be done by calculating a Global Fitness Score (GFS) based on performances attained and cardiovascular responses observed during physical exercises (3 min step test with measurement of heart rate and blood pressure, number of time subject can stand from a chair within 1 min., handgrip strength measure, "reach-test" to assess osteo-articular mobility of back and hips, balance test). Results obtained from this GFS will be compared to maximal power output calculated from a submaximal spirometry at 25, 50, 75 and 100 W M.

DETAILED DESCRIPTION:
Sedentarity is a risk factor for overweight, insulin resistance and diabetes mellitus. Several randomized clinical trials have shown that lifestyle interventions including exercise are efficient in improving metabolic homeostasis in overweight and obese patients. This may be related sedentarity being associated with low physical fitness, and to training enhancing it through multiple systems effects (cardiovascular and respiratory systems, central nervous system, osteo-articular system).

Although there is increasing evidence that low physical fitness is a risk factor for many non-communicable diseases, the early identification of subjects at risk remains inadequate due to the absence of clear anamnestic and clinical criteria. Defining physical fitness. For the same reason, the monitoring of subjects following lifestyle interventions remains suboptimal.

The aim of this study is to develop a simple field tool to non-invasively assess global physical fitness in overweight patients participating to a physical activity program.

Eigtheen male and female subjects, aged 18-50 years, BMI >27 kg/m2 referred to a physical activity intervention by their primary care physician, will be included. Their physical fitness will be assessed at inclusion (ie before starting the exercise program) and at the end of the 3-month program.This will be done by calculating a Global Fitness Score (GFS) based on performances attained and cardiovascular responses observed during 5 physical exercises (3 min step test with measurement of heart rate and blood pressure, number of time subject can stand from a chair within 1 min., handgrip strength measure, "reach-test" to assess osteo-articular mobility of back and hips, balance test). Results obtained from this GFS will be compared to maximal power output calculated from a submaximal spirometry at 25, 50, 75 and 100 W Primary outcome are: GFS (composite of a score of physical endurance, two scores of muscle strength, one score of balance, and one score of osteo-articular mobility) before and after 3 months of intervention.

Secondary outcomes are: physical activity questionnaire, maximal power output; maximal oxygen consumption; fat oxidation; fasting metabolic profile before and after 3 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI >27 kg/m2

Exclusion Criteria:

* cardio-respiratory diseases
* severe osteo-articular diseases
* any condition associated with contra-indication to exercise.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Overweight subjects referred to a physical activity intervention by their primary care physician
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Global Fitness Score before and after 3 months physical training | After 3 month physical training
  Global fitness score ranges between 0 (very low fitness) and 30 (optimal fitness). It is calculated as the sum of scores obtained with 5 simple field tests (Chester step test, score 0-10; handgrip, score 0-5; sit-and stand test, score 0-5; Sit and reach test, score 0-5; Flamingo test, score 0-5)

CONTACTS AND LOCATIONS:
Overall Officials: Charly Bulliard, MD, Study Chair — Hopital Intercantonal de la Broye, Estavayer le-lac, Switzerland
Locations (1):
- Hopital Intercantonal de la Broye, Estavayer-le-Lac, Canton of Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided